CLINICAL TRIAL: NCT06003036
Title: Accelerated Neuromodulation of Prefrontal Circuitry During Clozapine Treatment
Brief Title: Accelerated Transcranial Magnetic Stimulation for People With Schizophrenia Treated With Clozapine
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Deepak K. Sarpal, M.D. (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor-Investigator, Deepak K. Sarpal, M.D., Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: STUDY23050056; R21MH134128 (NIH)
Record Dates: First submitted 2023-08-08; First posted 2023-08-21 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Schizophrenia; Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- iTBS, then Sham (Experimental)
  Interventions: Device: sham stimulation; Device: transcranial magnetic stimulation
- Sham, then iTBS (Experimental)
  Interventions: Device: sham stimulation; Device: transcranial magnetic stimulation

INTERVENTIONS:
Device: sham stimulation — sham delivery of transcranial magnetic stimulation
Device: transcranial magnetic stimulation — accelerated intermittent theta burst stimulation

SUMMARY:
In this study, the investigators will examine whether a type of repetitive transcranial magnetic stimulation called accelerated intermittent theta burst stimulation (iTBS) can augment neurocognition in individuals who receive treatment with clozapine. Following a baseline evaluation and magnetic resonance imaging (MRI), participants will undergo a session of iTBS +MRI and session of sham delivery + MRI. The order for these sessions will be blinded and randomized. The investigators predict that accelerated iTBS will enhance neurocognition relative to sham delivery.

ELIGIBILITY:
Inclusion Criteria:

1. A current Diagnostic and Statistical Manual of Mental Disorders 5 (DSM 5)-defined diagnosis of schizophrenia or schizoaffective disorder
2. age 18-50 years
3. at least 4 months of clozapine treatment
4. history of at least 2 failed antipsychotic trials
5. competency and willingness to sign informed consent
6. A clinically optimized dosage of clozapine, unchanged for at least 1 month, with a minimum of 150 mg/day

Exclusion Criteria:

1. Serious neurologic or medical condition/treatment that impacts the brain
2. a significant risk of suicidal or homicidal behavior
3. cognitive or language limitations, or any other factor that would preclude subjects providing informed consent
4. pregnancy or postpartum (<6 weeks after delivery or miscarriage)
5. history of treatment with electroconvulsive therapy
6. contraindications for magnetic resonance imaging (e.g., a pacemaker)
7. Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders 5 (DSM 5)-verified moderate or severe substance use disorder, including alcohol use disorder
8. seizure disorder or prior history of seizures on clozapine
9. patients taking both bupropion and clozapine
10. prior issues with intermittent theta burst stimulation/transcranial magnetic stimulation administration

Concomitant treatment with serotonin and norepinephrine reuptake inhibitors will be examined on a case-by-case basis.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
change in brain functional connectivity within the prefrontal cortex | 1 hour
  Examine changes in left dorsolateral prefrontal cortex-basal forebrain functional connectivity following adjunctive accelerated intermittent theta burst stimulation (iTBS)
change in activation of the working memory network | 1 hour
  Examine whether accelerated intermittent theta burst stimulation (iTBS) is associated with functional magnetic resonance imaging (fMRI)-based changes in activation of the working memory network during AX-continuous performance task engagement

SECONDARY OUTCOMES:
explore change in functional magnetic resonance imaging (fMRI) measures versus plasma n-desmethylclozapine/clozapine ratios | 1 month
  In exploratory analyses we will compare change in dorsolateral prefrontal cortex-basal forebrain functional connectivity and change in working memory network activation in relation to plasma n-desmethylclozapine/clozapine ratios.

CONTACTS AND LOCATIONS:
Overall Officials: Deepak K Sarpal, M.D., Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Western Psychiatric Hospital/University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
de-identified individual participant data to the National Institute of Mental Health (NIMH) data archive